CLINICAL TRIAL: NCT04478513
Title: A Phase I, Open-label, Non-randomised Study to Assess the Effect of Fluvoxamine (CYP1A2 Inhibitor) and Smoking (CYP1A2 Inducer) on the Pharmacokinetics of a Single Oral Dosing of AZD4635 in Healthy Volunteers
Brief Title: A Study to Assess the Effect of Fluvoxamine and Smoking on Pharmacokinetics ( the Movement of Drugs Within the Body) of AZD4635 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8730C00007
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteer/DDI Study
Keywords: CYP1A2 Inhibitor; CYP1A2 Inducer; Pharmacokinetics; Adenosine 2A receptor (A2AR) antagonist
MeSH Terms: interventions — Fluvoxamine

STUDY DESIGN:
Intervention Model Description: The study is two-period, fixed sequence study in healthy volunteers who are either smokers or non-smokers. Twenty-eight subjects are planned to be enrolled; 14 subjects who are smokers and 14 subjects who are non-smokers. Enrolling 28 subjects will ensure that at least 12 subjects each from the smoking and the non-smoking populations are evaluated in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): Pre-specified group of participants.
  Interventions: Drug: AZD4635; Drug: Fluvoxamine
- Non-smokers (Experimental): Pre-specified group of participants.
  Interventions: Drug: AZD4635; Drug: Fluvoxamine

INTERVENTIONS:
Drug: AZD4635 — During each treatment period subjects will receive a single dose of AZD4635 under fasting conditions.
Drug: Fluvoxamine — Daily oral single doses of fluvoxamine are planned to be administered to healthy volunteers in Treatment Period 2.

SUMMARY:
This study is a Phase I, open-label, non-randomized, 2-period, fixed-sequence study in healthy volunteers who are either smokers or non-smokers, performed at a single Clinical Unit.

DETAILED DESCRIPTION:
The study will comprise:

* A screening period of up to 28 days;
* Two treatment periods lasting a total of 17 days from admission to the Clinical Unit (Day -1) to discharge (Day 16). During each treatment period subjects will receive a single dose of AZD4635 under fasting conditions. Period 1 is designed to evaluate the pharmacokinetics (PK) of AZD4635 in healthy smokers and non-smokers. Period 2 is designed to evaluate the effect of fluvoxamine on the PK of AZD4635 in healthy smokers and non-smokers.
* A follow-up call will take place between 6 to 9 days after the last dose of fluvoxamine, to ensure the well-being of the subjects. Completion of the last follow-up call or unscheduled follow-up visit will be considered the end of the study.

Each subject will be involved in the study for a maximum of 53 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects of non-childbearing potential subjects aged 18 - 55 years (inclusive at screening) with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18.5 and 32.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg, inclusive.
* Willingness and ability to comply with study and follow-up procedures.
* Subjects who are recruited as non-smokers should have no history of smoking cigarettes for >6 months and test negative for urine cotinine levels at screening and admission.
* Subjects who are recruited as smokers must have a history of smoking >10 cigarettes/day for >6 months and have urine cotinine levels over 500 ng/ml at screening and admission.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the principal investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of cardiac disease; concurrent electroconvulsive therapy, diabetes mellitus, epilepsy, bleeding disorders (especially GI bleeding), mania and susceptibility to angle-closure glaucoma.
* Presence of refractory nausea and vomiting or chronic GI diseases.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the PI (based on laboratory parameters).
* Any clinically significant abnormal findings in vital signs at screening as judged by the PI.
* Systolic blood pressure (BP) >140 and/or diastolic BP > 90 mmHg, or history of hypertension at screening.
* Any confirmed clinically significant abnormalities on 12-lead ECG at screening, as judged by the PI.
* Haemoglobin A1c (HbA1c) >5.7% at the screening visit.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibodies.
* Known or suspected history of drug abuse, within the past 2 years, as judged by the PI.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI.
* Positive screen for drugs of abuse at screening or admission to the study centre.
* Use of herbal preparations/medications within 14 days prior to the administration of the first dose of AZD4635.
* Subject who has had prescription or non-prescription drugs or other products known to be sensitive to Breast cancer resistance protein.
* Use of any prescribed or non prescribed medication including antacids, analgesics, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP.
* Subjects who have involvement with AstraZeneca or Parexel or are study site employee or their close relatives.
* Subjects who have previously been enrolled in this study or have previously received AZD4635.
* Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to infinity (AUC) | Days 1-6 and Days 11-16
  To assess the effect of fluvoxamine and smoking on the PK of AZD4635 following single oral dosing in healthy volunteers
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) | Days 1-6 and Days 11-16
  To assess the effect of fluvoxamine and smoking on the PK of AZD4635 following single oral dosing in healthy volunteers
Maximum observed plasma concentration (Cmax) | Days 1-6 and Days 11-16
  To assess the effect of fluvoxamine and smoking on the PK of AZD4635 following single oral dosing in healthy volunteers

SECONDARY OUTCOMES:
Number of subjects with adverse events, serious adverse events and deaths | From Screening upto Day 24
  To assess adverse events as a variable of safety and tolerability of AZD4635 when dosed with and without fluvoxamine in smokers and non-smokers

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, Dr., Principal Investigator — Parexel Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the
  Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home